CLINICAL TRIAL: NCT05122182
Title: An Investigator Initiated, International Multi-Centre, Multi-Arm, Multi-Stage Randomised Double Blind Placebo Controlled Trial of Angiotensin Receptor Blocker (ARB) & Chemokine Receptor Type 2 (CCR2) Antagonist for the Treatment of COVID-19
Brief Title: Controlled Trial of Angiotensin Receptor Blocker (ARB) & Chemokine Receptor Type 2 (CCR2) Antagonist for the Treatment of COVID-19
Acronym: CLARITY 2
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Withdrawal of funding support from the trial funder.
Sponsor: University of Sydney (Other)
Collaborators: The George Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CTC0312
Record Dates: First submitted 2021-11-14; First posted 2021-11-16 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: COVID-19; SARS-CoV2 Infection
Keywords: COVID-19; SARS-CoV2; Angiotensin Receptor Blocker (ARB); C-C chemokine receptor type 2 (CCR2) antagonist
MeSH Terms: conditions — COVID-19 | interventions — candesartan cilexetil; propagermanium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Interventional Arm (Experimental): Titratable candesartan with commencing dose 4mg tablets twice daily (daily dose 8 mg) + fixed dose repagermanium one x 120mg immediate release capsule twice daily (total daily dose 240mg). Treatment will continue for 28 days.
  Interventions: Drug: Candesartan Cilexetil; Drug: Repagermanium
- Control Arm #1 (Placebo Comparator): Titratable candesartan with commencing dose 4mg tablets twice daily (daily dose 8 mg) + matched placebo repagermanium one capsule twice daily. Treatment will continue for 28 days.
  Interventions: Drug: Candesartan Cilexetil; Drug: Repagermanium Placebo
- Control Arm #2 (Placebo Comparator): Titratable matched placebo candesartan one tablet twice daily + matched placebo repagermanium one capsule twice daily. Treatment will continue for 28 days.
  Interventions: Drug: Candesartan Placebo; Drug: Repagermanium Placebo

INTERVENTIONS:
Drug: Candesartan Cilexetil — Angiotensin Receptor Blocker (ARB)
  Arms: Control Arm #1; Interventional Arm
Drug: Repagermanium — C-C chemokine receptor type 2 (CCR2) antagonist
  Other Names: DMX-200
  Arms: Interventional Arm
Drug: Candesartan Placebo — Angiotensin Receptor Blocker (ARB) placebo
  Arms: Control Arm #2
Drug: Repagermanium Placebo — C-C chemokine receptor type 2 (CCR2) antagonist placebo
  Arms: Control Arm #1; Control Arm #2

SUMMARY:
CLARITY 2.0 is an investigator-initiated trial that will evaluate the safety and efficacy of dual treatment with repagermanium, a CCR2 antagonist, and candesartan, an ARB, in patients hospitalised with COVID-19 disease.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged ≥ 18 years (maximum 65 years old in India).
2. Laboratory-confirmed diagnosis of SARS-CoV-2 infection within 10 days prior to randomisation. (Confirmation must be through Reverse Transcription Polymerase Chain Reaction [RT-PCR] method)
3. Intended for hospital admission for management of COVID-19.
4. Patients with moderate (respiratory rate of ≥ 24/minute or SPO2: 90% to ≤ 93% on room air) or severe (respiratory rate of ≥ 30/minute or SPO2: <90% on room air) COVID-19.
5. Systolic Blood Pressure (SBP) ≥ 120 mmHg OR SBP ≥ 115 mmHg and currently treated with a non-RAASi BP lowering agent that can be ceased.
6. Willing and able to comply with all study requirements, including treatment, timing and/or nature of required assessments.
7. Documented informed consent.

Exclusion Criteria:

1. Currently treated with an ACEi, ARB or aldosterone antagonist, aliskiren, or ARNi
2. Intolerance of ARBs
3. Serum potassium >5.5 mmol/L
4. An estimated Glomerular Filtration Rate (eGFR) <30ml/min/1.732m
5. Known biliary obstruction, known severe hepatic impairment (Child-Pugh-Turcotte score 10-15)
6. Pregnancy, lactation, or inadequate contraception.
7. Participation in a study of a novel investigational product within 28 days prior to randomisation.
8. Plans to participate in another study of a novel investigational product during this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2022-01-07 (Actual); Primary Completion 2022-08-15 (Actual); Study Completion 2023-01-28 (Actual)

PRIMARY OUTCOMES:
Clinical Health Score at day 14 | 14 days
  The primary objective is to evaluate the safety and efficacy of dual treatment with repagermanium and candesartan in patients hospitalised with COVID-19 disease, assessed by the Clinical Health Score at day 14, which is determined within an 8-point ordinal scale of health status:
  1. Not hospitalised, no limitations on activities.
  2. Not hospitalised, limitation on activities.
  3. Hospitalised, not requiring supplemental oxygen.
  4. Hospitalised, requiring supplemental oxygen by mask or nasal prongs.
  5. Hospitalised, on non-invasive ventilation or high-flow oxygen devices.
  6. Hospitalised, requiring intubation and mechanical ventilation.
  7. Hospitalised, on invasive mechanical ventilation and additional organ support (ECMO).
  8. Death.

SECONDARY OUTCOMES:
Clinical Health Score at day 28 | 28 days
  The primary objective is to evaluate the safety and efficacy of dual treatment with repagermanium and candesartan in patients hospitalised with COVID-19 disease, assessed by the Clinical Health Score at day 28, which is determined within an 8-point ordinal scale of health status:
  1. Not hospitalised, no limitations on activities.
  2. Not hospitalised, limitation on activities.
  3. Hospitalised, not requiring supplemental oxygen.
  4. Hospitalised, requiring supplemental oxygen by mask or nasal prongs.
  5. Hospitalised, on non-invasive ventilation or high-flow oxygen devices.
  6. Hospitalised, requiring intubation and mechanical ventilation.
  7. Hospitalised, on invasive mechanical ventilation and additional organ support (ECMO).
  8. Death.
ICU admission | 28 days
  The secondary objectives are to evaluate the safety and efficacy of dual treatment with repagermanium and candesartan in patients hospitalised with COVID-19 disease, assessed by incidence of ICU admission in days 0-28.
Death | 28 days
  The secondary objectives are to evaluate the safety and efficacy of dual treatment with repagermanium and candesartan in patients hospitalised with COVID-19 disease, assessed by incidence of deaths in days 0-28.
Time to death | 28 days
  The secondary objectives are to evaluate the safety and efficacy of dual treatment with repagermanium and candesartan in patients hospitalised with COVID-19 disease, assessed from hospital admission to death.
Acute Kidney Injury | 28 days
  The secondary objectives are to evaluate the safety and efficacy of dual treatment with repagermanium and candesartan in patients hospitalised with COVID-19 disease, assessed by incidence of acute kidney injury in days 0-28.
Respiratory Failure | 28 days
  The secondary objectives are to evaluate the safety and efficacy of dual treatment with repagermanium and candesartan in patients hospitalised with COVID-19 disease, assessed by incidence of respiratory failure in days 0-28.
Length of hospital admission | 28 days
  The secondary objectives are to evaluate the safety and efficacy of dual treatment with repagermanium and candesartan in patients hospitalised with COVID-19 disease, assessed by days of inpatient stay from admission to discharge or death.
Length of ICU Admission | 28 days
  The secondary objectives are to evaluate the safety and efficacy of dual treatment with repagermanium and candesartan in patients hospitalised with COVID-19 disease, assessed by days in ICU from admission to transfer to ward or death.
Requirement of ventilatory support | 28 days
  The secondary objectives are to evaluate the safety and efficacy of dual treatment with repagermanium and candesartan in patients hospitalised with COVID-19 disease, assessed by count of days with ventilation in days 0-28.
Requirement of dialysis | 28 days
  The secondary objectives are to evaluate the safety and efficacy of dual treatment with repagermanium and candesartan in patients hospitalised with COVID-19 disease, assessed by count of days with dialysis in days 0-28.
Clinical Health Score at day 60 | 60 days
  The primary objective is to evaluate the safety and efficacy of dual treatment with repagermanium and candesartan in patients hospitalised with COVID-19 disease, assessed by the Clinical Health Score at day 60, which is determined within an 8-point ordinal scale of health status:
  1. Not hospitalised, no limitations on activities.
  2. Not hospitalised, limitation on activities.
  3. Hospitalised, not requiring supplemental oxygen.
  4. Hospitalised, requiring supplemental oxygen by mask or nasal prongs.
  5. Hospitalised, on non-invasive ventilation or high-flow oxygen devices.
  6. Hospitalised, requiring intubation and mechanical ventilation.
  7. Hospitalised, on invasive mechanical ventilation and additional organ support (ECMO).
  8. Death.
Clinical Health Score at day 90 | 90 days
  The primary objective is to evaluate the safety and efficacy of dual treatment with repagermanium and candesartan in patients hospitalised with COVID-19 disease, assessed by the Clinical Health Score at day 90, which is determined within an 8-point ordinal scale of health status:
  1. Not hospitalised, no limitations on activities.
  2. Not hospitalised, limitation on activities.
  3. Hospitalised, not requiring supplemental oxygen.
  4. Hospitalised, requiring supplemental oxygen by mask or nasal prongs.
  5. Hospitalised, on non-invasive ventilation or high-flow oxygen devices.
  6. Hospitalised, requiring intubation and mechanical ventilation.
  7. Hospitalised, on invasive mechanical ventilation and additional organ support (ECMO).
  8. Death.
Clinical Health Score at day 180 | 180 days
  The primary objective is to evaluate the safety and efficacy of dual treatment with repagermanium and candesartan in patients hospitalised with COVID-19 disease, assessed by the Clinical Health Score at day 180, which is determined within an 8-point ordinal scale of health status:
  1. Not hospitalised, no limitations on activities.
  2. Not hospitalised, limitation on activities.
  3. Hospitalised, not requiring supplemental oxygen.
  4. Hospitalised, requiring supplemental oxygen by mask or nasal prongs.
  5. Hospitalised, on non-invasive ventilation or high-flow oxygen devices.
  6. Hospitalised, requiring intubation and mechanical ventilation.
  7. Hospitalised, on invasive mechanical ventilation and additional organ support (ECMO).
  8. Death.

OTHER OUTCOMES:
Incidence of Hypotension | 28 days
  The specific safety objectives are to evaluate the safety of dual treatment with repagermanium and candesartan in patients hospitalised with COVID-19 disease, assessed by incidence of hypotension in days 0-28.
Incidence of Hyperkalemia | 28 days
  The specific safety objectives are to evaluate the safety of dual treatment with repagermanium and candesartan in patients hospitalised with COVID-19 disease, assessed by incidence of hyperkalemia in days 0-28.
Incidence of Deranged Liver Function Tests | 28 days
  The specific safety objectives are to evaluate the safety of dual treatment with repagermanium and candesartan in patients hospitalised with COVID-19 disease, assessed by incidence of deranged liver function tests in days 0-28.
Total Serious Adverse Events (SAEs) | 28 days
  The specific safety objectives are to evaluate the safety of dual treatment with repagermanium and candesartan in patients hospitalised with COVID-19 disease, assessed by total number of SAEs in days 0-28.
Incidence of hospital readmission | 90 days
  Admission for overnight stay up to day 90 following initial hospital discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Meg Jardine, Study Chair — NHMRC Clinical Trials Centre, The University of Sydney; Vivekanand Jha, Study Chair — The George Institute
Locations (10):
- India (10):
  - Jawaharlal Nehru Medical College and Hospital, Aligarh
  - Government Medical College and Hospital, Chandigarh
  - Samishta Hospital and Research Institute, Guntur
  - Maharaja Agrasen Hospital, Jaipur
  - Amrita Institute of Medical Science, Kochi
  - Kasturba Medical College, Mangaluru
  - DM Wayanad Institute of Medical Sciences, Meppādi
  - Sterling Hospital, Nigdi
  - Jivanrekha Multi-Speciality Hospital, Pune
  - All India Institute of Medical Sciences, Raipur, Raipur

IPD SHARING:
Plan to Share IPD: Yes
Trial data will be disseminated in the form of a publication to a relevant clinical journal and presentation at appropriate scientific conferences.
  Individual participant data that underlie the results reported, after de-identification (text, tables, figures, and appendices), may be shared with Investigators whose proposed use of the data has been approved by an independent review committee ("learned intermediary") identified for this purpose.
Supporting Information: Study Protocol, ICF, CSR
Access Criteria: Data will be available after publication for an indefinite time / for a finite time (specify dates) All data requests will be considered by the primary sponsor on a case-by-case basis. Requests must include a methodologically sound proposal. Specific conditions of use may apply and will be specified in a data sharing agreement that the requester must agree to before access is granted.
  Access can be requested via the Health Data Australia catalogue
URL: https://researchdata.edu.au/health/

REFERENCES:
- [Derived] O'Hara DV, Bassi A, Wilcox A, Jha V, Rathore V, D'Cruz S, Snelling TL, Jones M, Totterdell J, Bangi A, Jain MK, Pollock C, Burrell L, Fox G, Jones C, Kotwal S, Faridah Syed Omar S, Jardine M; CLARITY 2.0 trial investigators. Combination of the chemokine receptor type 2 (CCR2) antagonist DMX-200 and candesartan for COVID-19: a randomised controlled trial. BMJ Open. 2024 Oct 22;14(10):e081790. doi: 10.1136/bmjopen-2023-081790. PMID 39438096